CLINICAL TRIAL: NCT05801016
Title: Esplorare l'Effetto di un Protocollo Combinato di Realtà Virtuale e Autobiographical Recall su Memoria, Percezione, Affetto in Pazienti Con Anoressia Nervosa: Uno Studio Preliminare
Brief Title: Virtual Reality and Autobiographical Recall in Anorexia Nervosa: a Preliminary Study
Acronym: VIREC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 05C923
Record Dates: First submitted 2023-03-08; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anorexia nervosa (Other): Female anorexia nervosa patients
  Interventions: Behavioral: Emerging Technologies and Training in Neurosciences
- Healthy controls (Other): Healthy female control participants
  Interventions: Behavioral: Emerging Technologies and Training in Neurosciences

INTERVENTIONS:
Behavioral: Emerging Technologies and Training in Neurosciences — Combination of body-swapping technique, Virtual Reality Body Size estimation tasks and Autobiographic Recall

SUMMARY:
Clinical trial in patients with Anorexia Nervosa using body-swapping technique e Virtual Reality Body Size estimation tasks and Autobiographic Recall on sympton remission (EDI-3; EDE-Q), body satisfaction and perception

ELIGIBILITY:
Inclusion Criteria:

* Anorexia Nervosa
* Body mass index equal or superior to 15 kg/m2
* Mother tongue Italian
* Semiresidential rehabilitation program

Exclusion Criteria:

* Other eating disorders
* Neurological disorders , clinical history of cerebral damage, presence of psychiatric disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in estimation of body weight | At baseline and after 12 months
  Overestimation of body weight measured through Eating Disorder Inventory (EDI-3)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Riva, prof, Study Director — università cattolica Milano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No